CLINICAL TRIAL: NCT04374500
Title: The Effect of the Adipocyte-derived Hormone Leptin on Endothelial Function in Healthy Men and in Persons With Known Cardiovascular Disease
Brief Title: Leptin Infusion and Endothelial Vasomotor Response
Acronym: LIVARM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stefan Soderberg (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor-Investigator, Stefan Soderberg, Professor, Umeå University
Organization: Umeå University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 05-150M
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Results first posted 2020-07-17 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-07

CONDITIONS: Endothelial Dysfunction; Obesity; Vasodilation; Venous Occlusion Plethysmography
MeSH Terms: conditions — Obesity; Aneurysm | interventions — Vasodilator Agents; Bradykinin; Acetylcholine; Nitroprusside; Verapamil; Substance P; Single Person

STUDY DESIGN:
Intervention Model Description: In protocol 1, each participant was examined once. Leptin was given intraarterially in the forearm in increasing doses and forearm blood flow (FBF) was measured. No masking, no randomisation.
  In protocol 2, each participant was examined twice and they got either leptin or saline intraarterially in the forearm at least 2 weeks apart, and the order was randomised. Concomitantly, they got four vasodilatators (bradykinin, acetylcholine, sodium nitroprusside and verapamil) intraarterially in a randomised order.
  In protocol 3, each participant was examined once and the three vasodilatators (substance P, acetylcholine, and sodium nitroprusside) were given intraarterially in the forearm in a randomised order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Leptin infusion (Experimental): This applies to protocol 1 when 10 healthy men got leptin infused locally in the forearm and forearm blood flow (FBF) was measured. The other forearm was used as the control.
  Interventions: Drug: Leptin infusion in healthy men
- Leptin infusion plus vasodilator infusion (Experimental): This applies to protocol 2 when 10 healthy men got either a background infusion of leptin or saline locally in the forearm when measuring vasoresponse (FBF) to four vasodilatators. Each participant had two examinations with either leptin or saline and the order was randomised. The other forearm was used as the control.
  Interventions: Drug: Leptin infusion plus vasodilators in healthy men
- Vasodilator infusion in CAD patients (Experimental): This applies to protocol 3 when 83 men and women with known CAD (coronary artery disease) got three vasodilators locally infused in the forearm while measuring vasoresponse (FBF). The other forearm was used as the control.
  Interventions: Drug: Vasodilators in CAD patients

INTERVENTIONS:
Drug: Leptin infusion plus vasodilators in healthy men — This applies only to protocol 2 with two arms (leptin or saline) where four vasodilatators (bradykinin, acetylcholine, sodium nitroprusside and verapamil) were infused concomitantly
  Other Names: Four vasodilators (bradykinin, acetylcholine, sodium nitroprusside and verapamil) on top of leptin or saline infusion
  Arms: Leptin infusion plus vasodilator infusion
Drug: Leptin infusion in healthy men — This applies only to protocol 1 when only leptin was given
  Other Names: Leptin infusion only and blood flow measured
  Arms: Leptin infusion
Drug: Vasodilators in CAD patients — This applies only to protocol 3
  Other Names: Three vasodilators (acetylcholine, sodium nitroprusside, substance P) only, related to endogenous leptin levels
  Arms: Vasodilator infusion in CAD patients

SUMMARY:
Adipose tissue is an active endocrine organ producing several hormones with circulatory and metabolic effects. In 1994, the hormone leptin was discovered. The lack of this hormone explained extreme obesity in rare patients and parenteral substitution restored body weight and metabolic disturbances. It was however soon discovered that most humans had too high levels which were related to development of cardiovascular diseases and diabetes. It was hypothesised that leptin induced vessel dysfunction which could explain this association.

In this study, we wanted to examine the association between leptin and vessel function by using the venous occlusion plethysmography method. We used three protocols to evaluate this association.

First protocol. In ten healthy males, leptin was infused locally in the forearm and forearm blood flow (FBF) was measured.

Second protocol. In ten healthy males, leptin or normal saline was infused locally in the forearm and FBF was measured. Concomitantly, four vasodilatators were infused locally in the forearm in a randomised order and the response (blood flow and fibrinolysis) was measured.

Third protocol. In eighty-three patients with known coronary artery disease, three vasodilators were infused locally in the forearm in a random order and response (FBF and fibrinolysis) was measured. The response was related to endogenous leptin levels.

The two first protocols were performed in Umeå, Sweden whereas the third was performed in Edinburgh, UK, all in 2006.

DETAILED DESCRIPTION:
Introduction High BMI and particularly fat mass index are associated with increased risk of coronary artery disease and other cardiovascular conditions, but the underlying mechanisms are not well understood. Endothelial dysfunction precedes atherosclerosis and represents an important link between obesity and cardiovascular events.

The adipose tissue produces cytokines and hormones (adipokines), which, in excess, may promote cardiovascular disease by proinflammatory, prothrombotic, dyslipidemic and atherosclerotic effects.

Leptin is an adipokine with pleiotropic effects and circulating leptin levels are positively associated with the amount of body fat. High plasma leptin levels (hyperleptinemia) associate with the development of atherosclerosis, hypertension and coronary artery disease (CAD). Leptin activates specific leptin receptors expressed, among other tissues, in vascular cells, suggesting that leptin may participate in the development of endothelial dysfunction and atherosclerosis.

However, the net effect of leptin on vasomotor function remains unclear, as both vasodilation and vasoconstriction have been reported. Leptin induces release of nitric oxide (NO) in vitro and elicits endothelium-dependent vasodilation in mice by inducing endothelial expression of NO synthase. In addition, studies in humans have shown that leptin infusion exerts vasodilatation. In contrast, others have shown leptin-induced vasoconstriction in vitro and impaired vasodilatation in dogs. Different mechanisms have been proposed causing increased peripheral vascular resistance, such as vascular inflammation, increased sympathetic nervous system (SNS) activity, increased endothelin-1 (ET-1) production, and decreased nitric oxide (NO) bioavailability.

Hyperleptinemia has been associated to states of altered fibrinolysis, which is common in diabetes, cardiovascular disease and obesity. However, whether leptin directly influences the endogenous fibrinolytic function remains unclear.

The aim of these studies was to evaluate the role of leptin on endothelial function in humans. For this purpose, the vasomotor and the fibrinolytic functions were assessed in healthy men during a state of pharmacologically induced hyperleptinemia. In a parallel study, the endothelial function was assessed in patients with established CAD and related to plasma leptin levels.

Material and Methods

Subjects Twenty healthy non-smoking male volunteers not taking any regular medication were recruited in Umeå, Sweden. 2). Eighty-three patients with established CAD were recruited from the cardiology outpatient clinic at the Royal Infirmary, Edinburgh, Scotland, and the characteristics of this cohort have been reported previously. These patients had stable angina and had a prior angiographic documentation of ≥50% luminal stenosis of at least one major epicardial coronary vessel. Written informed consent was obtained from each subject and the studies were carried out in accordance with the Declaration of Helsinki.

Venous occlusion plethysmography Subjects abstained from alcohol for 24 hours and from food, tobacco and caffeine-containing drinks for at least 4 hours before each study visit. All studies were carried out in a quiet temperature-controlled room maintained at 22-25 degrees Celsius (ºC). A 17-G venous cannula was inserted into the antecubital vein of each arm and the brachial artery of the non-dominant arm was cannulated with a 27-G needle (Cooper's Needle Works Ltd, UK). Bilateral forearm blood flow (FBF) was measured by venous occlusion plethysmography using mercury-in-silastic strain gauges. Blood pressure and heart rate were measured using a semi-automated non-invasive sphygmomanometer. To avoid acute vasomotor effects, all medications were withheld on the morning of each study.

Study design

Protocol 1 In ten healthy male volunteers, recombinant human leptin (Sigma-Aldrich, Saint-Louis, Missouri, USA) was infused intra-arterially at ascending doses of 80, 800 and 8,000 ng/min (6 minutes each). Heart rate, blood pressure, FBF, leptin, tissue plasminogen activator (tPA) antigen and plasminogen activator inhibitor type 1(PAI-1) antigen concentrations were determined at the end of each dose.

Protocol 2 In a double-blind randomized crossover study, ten healthy male volunteers received intra-arterial infusions of either leptin (800 ng/min) or saline on two separate occasions with at least 2 weeks between visits. FBF was measured in the infused and non-infused arms at baseline and at regular intervals during the one-hour leptin/saline infusion. Thereafter four vasodilators were infused concomitantly with intra-arterial leptin/saline infusions; bradykinin (endothelium-dependent vasodilator that releases tPA) at 100, 300 and 1,000 pmol/min (Clinalfa Ltd, Switzerland), acetylcholine (endothelium-dependent vasodilator that does not release tPA) at 5, 10 and 20 µg/min (Clinalfa Ltd, Switzerland), sodium nitroprusside (endothelium-independent vasodilator) at 2, 4 and 8 µg/min (David Bull laboratories, UK) and verapamil (endothelium-independent vasodilator) at 10, 30, 100 µg/min (Abbott UK Ltd) for 6 minutes at each concentration. Vasodilators were infused in a randomized order with a 15-minute saline washout period between each drug. Verapamil was always administered at the end because of its long-lasting vasomotor effects.

Venous blood was obtained from the infused and non-infused arms at baseline, before and during infusion of bradykinin, at 60 minutes and at the end of the study protocol.

Protocol 3 In patients with CAD (n=83), bilateral FBF was measured before and during intra-arterial infusions of substance P (endothelium-dependent vasodilator that releases tPA) at 2, 4 and 8 pmol/min (Clinalfa Ltd, Switzerland), acetylcholine at 5, 10 and 20 µg/min (as above) and sodium nitroprusside at 2, 4 and 8 µg/min (as above) for 6 minutes at each concentration. Bradykinin was not administered because many subjects were being treated with angiotensin-converting enzyme inhibition and this markedly potentiates its vasodilator and fibrinolytic effects. The vasodilators were administered in a randomized order with a 15-minute saline washout period between each drug. Venous blood samples were obtained before and during intra-arterial infusion of substance P to measure fibrinolytic markers.

Venous Sampling and Assays Fasting venous blood samples were drawn into tubes containing acidified buffered citrate or trisodium citrate. Samples were collected immediately onto ice and centrifuged at 2,000 g for 30 min. Platelet-free plasma and serum were stored at -80°C before assay. Brain natriuretic peptide (BNP), cholesterol and glucose concentrations were determined according to clinical routine, and high sensitivity C-reactive protein (hsCRP) with a highly sensitive assay using particle-enhanced immunonephelometry (Behring BN II nephelometer). Plasma leptin concentrations were measured using a double-antibody radioimmunoassay (Millipore, Billerica, Massachusetts, USA). According to the literature, intra- and inter-assay coefficients of variation should be less than 5% at both low (2-4 ng/mL) and high (10-15 ng/mL) leptin concentrations. Plasma tPA and PAI-1 antigen concentrations were determined using enzyme-linked immunosorbent assays (Coaliza®, Chromogenix Ltd) and plasma tPA activity using a photometric method (Coatest tPA, Chromogenix Ltd). According to the manufacture, the coefficients of variation for fibrinolytic assays are 5.9% and 12% for tPA antigen and activity respectively, and 6.2% for PAI-1 antigen. Estimated net release of tPA (antigen and activity) was calculated as previously described after each dose of bradykinin or substance P, as the product of the infused forearm plasma flow and the difference in plasma levels between the infused and non-infused forearms.

ELIGIBILITY:
Inclusion criteria protocol 1 and 2;

* Healthy male
* No regular medication
* Non-smoking
* Abstain from alcohol for 24 hours and from food, tobacco and caffeine-containing drinks for at least 4 hours before each study visit

Inclusion criteria protocol 3;

* Established coronary artery disease
* Stable angina pectoris
* Documented ≥ 50% stenosis of at least one major epicardial coronary vessel

Exclusion criteria protocol 3;

* Coronary revascularisation within three months
* Diabetes mellitus
* Cardiac failure (ejection fraction <35% or New York Heart Association (NYHA) ≥2)
* Renal impairment (creatinine ≥200 µmol/L)
* Systolic blood pressure <100 or >190 mmHg

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only males chosen for protocol 1 and 2. The reason is that men are more easily cannulated in the forearm artery with less risk for vasospasm.
Enrollment: 103 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2006-10-27 (Actual); Study Completion 2006-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Söderberg, MD, PhD, Principal Investigator — Umeå University, Umeå Sweden
Locations (2):
- Umeå University Hopsital, Umeå, Sweden
- British Heart Foundation Centre for Cardiovascular Science, University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request, data can be shared.
Supporting Information: Study Protocol, ICF
Time Frame: On reasonable request
Access Criteria: Contact with principal investigator (email)

REFERENCES:
- [Derived] Gonzalez M, Robinson S, Mills NL, Eriksson M, Sandstrom T, Newby DE, Olsson T, Blomberg A, Soderberg S. Vasomotor and fibrinolytic effects of leptin in man. Scand Cardiovasc J. 2025 Dec;59(1):2478867. doi: 10.1080/14017431.2025.2478867. Epub 2025 Mar 19. PMID 40066842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty (20) healthy non-smoking male volunteers not taking any regular medication were recruited in Umeå, Sweden, ten (10) participated in protocol 1 and ten (10) in protocol 2.
  Eighty-three (83) men and women with established coronary artery disease were recruited from the cardiology outpatient clinic at the Royal Infirmary, Edinburgh, Scotland.
Pre-assignment Details: Protocol 1 and 2 were performed in Umeå, Sweden. The two protocols were separated in time (approximately 6 months). The total number of participants were 10+10 men, with altogether 30 examinations (protocol 1 - examined once and protocol 2 - examined twice). Protocol 3 was performed in UK, and 83 participants were examined once. Thus 103 participants with 113 examinations.
Groups:
- Leptin Infusion in Healthy Men: This applies to protocol 1 when 10 healthy men got infusion of leptin locally and forearm blood flow was measured with the other arm as the control.
- Leptin or Saline Infusion Plus Vasodilators in Healthy Men: This applies to protocol 2 when 10 healthy men got either a background infusion of leptin or saline when measuring vasoresponse to four vasodilatators. Each participant had two examinations with either leptin or saline and the order was randomised.
- Vasodilators in CAD Patients: This applies to protocol 3 when blood flow was measured in the forearm after infusion of 3 vasodilators, and leptin was not infused
Period: Overall Study
Arm/Group | Leptin Infusion in Healthy Men | Leptin or Saline Infusion Plus Vasodilators in Healthy Men | Vasodilators in CAD Patients
Started (Recruitment and study procedures in all protocols were performed in 2006) | 10 | 10 | 83
Completed | 10 (10 men completed the study.) | 10 (10 men completed 20 examinations.) | 83 (83 men and women competed 83 examinations.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Altogether 103 persons were investigated; 20 healthy males (10 in protocol - 1 examined once and 10 in protocol 2 - examined twice), and 83 men and women with CAD in protocol 3 (examined once). Thus altogether 113 examinations in 103 participants.
  As the participants in protocol 1 and 2 were recruited from a homogeneous group (healthy male students in Umeå, Sweden), baseline data ar given for protocol 1 and 2 combined.
Groups:
- Healthy Males and CAD Patients: Arm 1: Healthy males (n=10). Leptin was infused intra-arterially (IA) at ascending doses of 80, 800 and 8,000 ng/min. Bilateral forearm blood flow (FBF), heart rate, blood pressure, leptin, tissue plasminogen activator (tPA) antigen were determined.
  Arm 2: Healthy males (n=10). Leptin (800 ng/min) or saline was given IA with at least 2 weeks between visits. Vasodilators were infused concomitantly with IA leptin/saline infusions; bradykinin at 100, 300 and 1,000 pmol/min, acetylcholine (AcCh) at 5, 10 and 20 µg/min, sodium nitroprusside (SNP) at 2, 4 and 8 µg/min and verapamil at 10, 30, 100 µg/min, for 6 minutes at each concentration. Bilateral FBF, heart rate, blood pressure, leptin, tPA antigen were determined.
  Arm 3: CAD patients (n=83). IA infusions of substance P at 2, 4 and 8 pmol/min, AcCh at 5, 10 and 20 µg/min, and SNP at 2, 4 and 8 µg/min were given. Bilateral FBF, heart rate, blood pressure, leptin, tPA antigen were determined.
Arm/Group | Healthy Males and CAD Patients
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Mean (SD) are given for age at baseline examination for 20 healthy males in protocol 1 and 2, and for 83 men and women with CAD in protocol 3.
  Years
    Healthy males: number analyzed (Participants) | 20
    Healthy males | 26.4 (5.8)
    Coronary artery disease (CAD) patients: number analyzed (Participants) | 83
    Coronary artery disease (CAD) patients | 60 (6)
Sex: Female, Male [Count of Participants; unit: Participants] — Altogether 20 healthy males were studied in protocol 1 and 2, and 66 men and 17 women with CAD in protocol 3.
  Participants
    Female | 17
    Male | 86
Region of Enrollment [Count of Participants; unit: Participants] — Population: Protocol 1 and 2 was performed in Sweden, 10 participants and 30 examinations.
  Participants
    United Kingdom: number analyzed (Participants) | 83
    United Kingdom | 83
    Sweden: number analyzed (Participants) | 20
    Sweden | 20
tPA antigen [Mean (Standard Deviation); unit: ng/mL] — Population: Mean (SD) are given for baseline examination for 20 healthy males in protocol 1 and 2, and for 83 men and women with CAD in protocol 3.
  ng/mL
    Healthy males: number analyzed (Participants) | 20
    Healthy males | 9.0 (6.0)
    Coronary artery disease (CAD) patients: number analyzed (Participants) | 83
    Coronary artery disease (CAD) patients | 11.6 (4.5)
Leptin [Mean (Standard Deviation); unit: ng/mL] — Venous sample before infusion of leptin. Population: Mean (SD) are given for baseline examination for 20 healthy males in protocol 1 and 2, and for 83 men and women with CAD in protocol 3.
  ng/mL
    Healthy males: number analyzed (Participants) | 20
    Healthy males | 4.7 (3.6)
    Coronary artery disease (CAD) patients: number analyzed (Participants) | 83
    Coronary artery disease (CAD) patients | 13.2 (7.5)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — In all protocols, blood pressure (mmHg) was measured concomitantly using a semi-automated non-invasive sphygmomanometer. Population: Mean (SD) are given for baseline examination for 20 healthy males in protocol 1 and 2, and for 83 men and women with CAD in protocol 3.
  mmHg
    Healthy males: number analyzed (Participants) | 20
    Healthy males | 139 (14.2)
    Coronary artery disease (CAD) patients: number analyzed (Participants) | 83
    Coronary artery disease (CAD) patients | 130 (18)
Heart rate [Mean (Standard Deviation); unit: Beats per minute (SEM)] — Population: Mean (SD) are given for baseline examination for 20 healthy males in protocol 1 and 2, and for 83 men and women with CAD in protocol 3.
  Beats per minute (SEM)
    Healthy males: number analyzed (Participants) | 20
    Healthy males | 56 (5.9)
    Coronary artery disease (CAD) patients: number analyzed (Participants) | 83
    Coronary artery disease (CAD) patients | 57 (11)

OUTCOME MEASURES:

1. Primary Outcome: Forearm Blood-flow (FBF)
Description: The primary outcome in all protocols were local blood-flow in the forearm (FBF). This was measured by venous occlusion plethysmography using mercury-in-silastic strain gauges and the unit is mL/100mL of tissue/min. In protocol 1, the FBF response to increasing levels of leptin was evaluated, In protocol 2, the FBF response to vasodilators on top of leptin or saline infusion was evaluated, and in protocol 3, FBF was measured after infusion of vasodilators and no leptin was given.
Time Frame: 18 minutes in protocol 1, 3 hours in protocol 2, non-applicable (NA) in protocol 3
Measure: Mean (Standard Error); unit: ml/100 mg tissue/min
Groups:
- Leptin Infusion, no Saline Given: In protocol 1, leptin was infused and blood-flow (FBF) was measured.
- Leptin Plus Vasodilators: In protocol 2, leptin or saline was infused in the forearm which was followed by infusion of vasodilators. Blood flow (FBF) was measured.
- Vasodilators in CAD Patients: Blood flow was measured locally in the forearm (FBF) after infusion of vasodilators. No leptin was given.
Arm/Group | Leptin Infusion, no Saline Given | Leptin Plus Vasodilators | Vasodilators in CAD Patients
Number analyzed (Participants) | 10 | 10 | 83
ml/100 mg tissue/min
  Leptin infused | 1.75 (0.14) | 3.1 (0.4) | NA (NA) — Leptin not infused.
  Saline infused | NA (NA) — Saline not infused | 3.4 (0.4) | NA (NA) — Saline not infused

2. Secondary Outcome: Release of Fibrinolytic Variables (Tissue Plasminogen Activator [tPA] and Plasminogen Activator Inhibitor-1 [PAI-1])
Description: In all protocols, fibrinolytic variables were measured. In protocol 2 and 3, in the infused forearm after vasodilatation with bradykinin or substance P, respectively.
  The fibrinolytic variable measured in all protocols was tPA activity (IU/mL) and is reported here after the leptin infusion, when applicable.
Time Frame: 18 minutes in protocol 1, 3 hours in protocol 2, NA in protocol 3
Measure: Mean (Standard Error); unit: IU/mL
Groups:
- Leptin Infusion: In protocol 1, leptin was infused and the fibrinolytic variable tPA activity was measured.
- Leptin Plus Vasodilators: In protocol 2, leptin or saline was infused in the forearm which was followed by infusion of vasodilators. The fibrinolytic variable tPA activity was measured.
- Vasodilators in CAD Patients: The fibrinolytic variable tPA activity was measured in the forearm after infusion of vasodilators. No leptin was given.
Arm/Group | Leptin Infusion | Leptin Plus Vasodilators | Vasodilators in CAD Patients
Number analyzed (Participants) | 10 | 10 | 83
IU/mL
  Leptin infused | 0.56 (0.12) | 0.91 (0.38) | NA (NA) — Leptin not infused
  Saline infused | NA (NA) — Saline not infused | 0.73 (0.26) | NA (NA) — Saline not infused

3. Secondary Outcome: Leptin
Description: Plasma leptin concentration (ng/mL) was measured in all protocols, and in protocol 1 and 2, specifically in both infused and in non-infused arms. Data given are leptin concentrations in the infused arm at the end of the infusion.
Time Frame: 18 minutes in protocol 1, 3 hours in protocol 2, NA in protocol 3
Population: In arm 3, the participants were not given any leptin, endogenous leptin was measured
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Leptin Infusion: In protocol 1, blood flow in the infused forearm did not change with leptin infusion
- Leptin Plus Vasodilators: In protocol 2, blood flow in the infused forearm did not change with leptin infusion whereas blod flow changed as expected with vasodilators, but blunted with concomitant leptin infusion versus saline infusion
- Vasodilators in CAD Patients: Blood flow was measured locally in the forearm after infusion of vasodilators. No leptin was given.
Arm/Group | Leptin Infusion | Leptin Plus Vasodilators | Vasodilators in CAD Patients
Number analyzed (Participants) | 10 | 10 | 83
ng/mL
  Leptin infused | 186.2 (10.2) | 13.1 (3.4) | NA (NA) — Leptin was not infused
  Saline infused | NA (NA) — Saline not infused | 3.4 (1.2) | NA (NA) — Saline not infused

4. Secondary Outcome: Systolic Blood Pressure
Description: In all protocols, blood pressure (mmHg) was measured concomitantly using a semi-automated non-invasive sphygmomanometer. Systolic blood pressure is reported here after leptin or saline infusion, when applicable.
Time Frame: 18 minutes in protocol 1, 3 hours in protocol 2, NA in protocol 3
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Leptin Infusion in Healthy Men: In protocol 1, leptin was infused locally, and systolic blood pressure was measured.
- Leptin or Saline Infusion Plus Vasodilators in Healthy Men: In protocol 2, leptin or saline was infused in the forearm which was followed by infusion of vasodilators. Systolic blood pressure was measured simultaneously.
- Vasodilators in CAD Patients: Systolic blood pressure was not measured.
Arm/Group | Leptin Infusion in Healthy Men | Leptin or Saline Infusion Plus Vasodilators in Healthy Men | Vasodilators in CAD Patients
Number analyzed (Participants) | 10 | 10 | 83
mmHg
  Leptin infused | 140 (3.7) | 134 (3.3) | NA (NA) — Leptin was not infused
  Saline infused | NA (NA) — Saline not infused | 136 (2.9) | NA (NA) — Saline not infused

5. Secondary Outcome: Heart Rate
Description: In all protocols, heart rate (beats per minute) was measured concomitantly. Heart rate is reported here after leptin or saline infusion, when applicable.
Time Frame: 18 minutes in protocol 1, 3 hours in protocol 2, NA in protocol 3
Measure: Mean (Standard Error); unit: Beats per minute
Groups:
- Leptin Infusion in Healthy Men: In protocol 1, leptin was infused locally, and pulse rate was measured.
- Leptin or Saline Infusion Plus Vasodilators in Healthy Men: In protocol 2, leptin or saline was infused in the forearm which was followed by infusion of vasodilators. Pulse rate was measured simultaneously.
- Vasodilators in CAD Patients: Vasodilators were given locally but pulse rate was not measured.
Arm/Group | Leptin Infusion in Healthy Men | Leptin or Saline Infusion Plus Vasodilators in Healthy Men | Vasodilators in CAD Patients
Number analyzed (Participants) | 10 | 10 | 83
Beats per minute
  Leptin infused | 59 (1.5) | 66 (3.6) | NA (NA) — Leptin not infused
  Saline infused | NA (NA) — Saline not infused | 66 (2.6) | NA (NA) — Saline not infused

ADVERSE EVENTS:
Time Frame: During the actual infusion plus 24 hours.
Description: We measured blood pressure and pulse during and after the infusion and each participant was interrogated about subjective side effects like nausea, flush etc.
Groups:
- Leptin Infusion: In protocol 1, each participant got leptin locally in the studied forearm whereas the other forearm acted as control.
  No adverse effects were reported.
- Leptin Infusion Plus Vasodilator Infusion: In protocol 2, each participant got ether saline or leptin locally in the studied forearm whereas the other arm acted as control. Local vasodilators were given in the studied forearm on top of leptin/saline infusion. The experiment was repeated and each participant participated twice.
  No adverse effects were reported during leptin infusion.
- Saline Infusion Plus Vasodilator Infusion: In protocol 2, each participant got ether saline or leptin locally in the studied forearm whereas the other arm acted as control. Local vasodilators were given in the studied forearm on top of leptin/saline infusion. The experiment was repeated and each participant participated twice.
  No adverse effects were reported during saline infusion.
- Vasodilator Infusion in CAD Patients: In protocol 3, only vasodilators were given in the studied forearm, and no leptin was given.
  No adverse effects were reported.
Arm/Group | Leptin Infusion | Leptin Infusion Plus Vasodilator Infusion | Saline Infusion Plus Vasodilator Infusion | Vasodilator Infusion in CAD Patients
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/83
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/83

LIMITATIONS AND CAVEATS:
Sympathetic activity should have been measured simultaneously, but was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes